CLINICAL TRIAL: NCT03580694
Title: A Phase 1 Study of REGN4659 (Anti-CTLA-4 mAb) in Combination With Cemiplimab (Anti-PD-1 mAb) in the Treatment of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of REGN4659 in Combination With Cemiplimab in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Program reprioritization
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4659-ONC-1795
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; NSCLC; Anti-PD-1; Anti-CTLA-4; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cemiplimab Monotherapy (Experimental): In a single dose escalation cohort, participants will receive cemiplimab alone.
  Interventions: Drug: Cemiplimab
- Combination Therapy (Experimental): Dose Escalation cohorts:
  In 3 dose escalation cohorts, participants will receive a lead-in dose of REGN4659 followed by REGN4659 and cemiplimab in combination.
  In 4 dose escalation cohorts, participants will receive REGN4659 with cemiplimab in combination.
  Dose Expansion cohorts:
  In dose expansion cohorts, participants will receive combination regimens of REGN4659 and cemiplimab.
  Interventions: Drug: REGN4659; Drug: Cemiplimab

INTERVENTIONS:
Drug: REGN4659 — REGN4659 will be administered by intravenous (IV) infusion.
  Arms: Combination Therapy
Drug: Cemiplimab — Cemiplimab will be administered by intravenous (IV) infusion.
  Other Names: REGN2810

SUMMARY:
The objective of this trial is to study REGN4659 and cemiplimab in treatment-experienced, non-small cell lung cancer (NSCLC) patients. There are 2 phases of this study: a dose escalation phase and a dose expansion phase.

ELIGIBILITY:
KEY Inclusion Criteria:

1. Patients with histologically or cytologically documented squamous or non-squamous NSCLC with unresectable stage IIIB or stage IV disease
2. Combination dose escalation cohorts: Treatment-experienced patients who have received no more than 3 lines of systemic therapy including no more than 2 lines of cytotoxic chemotherapy, and for whom no available therapy has a high probability to convey clinical benefit.
3. Dose escalation cohort C: Anti-PD-1/PD-L1 naïve patients who have received 1 to 2 prior lines of cytotoxic chemotherapy including a platinum doublet-containing regimen
4. Expansion cohort(s): Anti-PD-1/PD-L1 experienced patients who have progressed while receiving therapy or within 6 months of stopping therapy for stage III or IV disease. Patients must not have permanently discontinued anti-PD-1/PD-L1 therapy due to treatment related AE. Patients must have received one line of anti-PD--1/PD-L1 immunotherapy. Patients may also have received one line of chemotherapy

KEY Exclusion Criteria:

1. Expansion cohort(s) only: Patients who have never smoked, defined as smoking ≤100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression. Patients are eligible if central nervous system (CNS) metastases are adequately treated and patients have neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. Patients must be off (immunosuppressive doses of) corticosteroid therapy
3. Expansion cohort(s) only: Patients with tumors tested positive for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) gene mutations or ROS1 fusions.
4. Radiation therapy within 2 weeks prior to enrollment and not recovered to baseline from any AE due to radiation
5. Patients who received prior treatment with an anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody
6. Previous treatment with idelalisib (ZYDELIG®) at any time

Note: Other protocol defined inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) during the dose escalation phase | Up to week 126
Rate of treatment emergent adverse events (TEAEs) | Up to week 126
Rate of immune-related adverse events (irAEs) | Up to week 126
Rate of serious adverse events (SAEs) | Up to week 126
Rate of deaths | Up to week 126
Laboratory abnormalities (grade 3 or higher per Common Terminology Criteria for Adverse Events [CTCAE]) | Up to week 126
Objective Response Rate (ORR) based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 during the dose expansion phase | Up to week 126
REGN4659 and cemiplimab concentrations in serum over time | Up to week 126

SECONDARY OUTCOMES:
ORR based on RECIST 1.1 during the dose escalation phase | Up to week 126
ORR based on immune-based therapy Response Evaluation Criteria (iRECIST) | Up to week 126
Best overall response (BOR) | Up to week 126
Duration of response (DOR) | Up to week 126
Disease control rate | Up to week 126
Progression-free-survival (PFS) based on RECIST 1.1 | Up to week 126
PFS based on iRECIST | Up to week 126
Overall survival (OS) | Up to week 126

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (6):
- United States (6):
  - Regeneron Investigational Site, Chicago, Illinois
  - Regeneron Investigational Site, Grand Rapids, Michigan
  - Regeneron Investigational Site, Charlotte, North Carolina
  - Regeneron Investigational Site, Oklahoma City, Oklahoma
  - Regeneron Investigational Site, Nashville, Tennessee
  - Regeneron Investigational Site, San Antonio, Texas